CLINICAL TRIAL: NCT05417945
Title: A Prospective, Multicenter, Single-group Target Value Clinical Study to Evaluate the Safety and Efficacy of JensClip Transcatheter Valve Repair System in the Treatment of Moderate to Severe Degenerative Mitral Regurgitation
Brief Title: A Prospective, Multicenter Study to Evaluate the JensClip Transcatheter Valve Repair System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jenscare Scientific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-2021-06
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Degenerative Mitral Valve Disease; Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JensClip transcatheter valve repair system (Experimental): Using the JensClip transcatheter valve repair system for the treatment of patients with moderate-severe or severe degenerative mitral regurgitation who are at high surgical risk.
  Interventions: Device: JensClip transcatheter valve repair system

INTERVENTIONS:
Device: JensClip transcatheter valve repair system — Transcatheter mitral valve repair system is derived from the "Edge-to-Edge" technique in traditional surgery. The principle is roughly to clamp the midpoint of the anterior leaflet and the midpoint of the posterior leaflet of the mitral valve to form a double-hole inflow channel and then improve the regurgitation.

SUMMARY:
The clinical trial study is designed as a prospective, multicenter, single-group target value clinical study to evaluate the safety and efficacy of the clinical investigational product and to evaluate its performance using the above clinical trial primary endpoint and secondary endpoint indicators.

DETAILED DESCRIPTION:
Transcatheter mitral valve repair system is derived from the "Edge-to-Edge" technique in traditional surgery. The principle is roughly to clamp the midpoint of the anterior leaflet and the midpoint of the posterior leaflet of the mitral valve to form a double-hole inflow channel and then improve the regurgitation.Using the JensClip transcatheter valve repair system for the treatment of patients with moderate-severe or severe degenerative mitral regurgitation who are at high surgical risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Echocardiographically confirmed moderate-severe or severe degenerative mitral regurgitation (regurgitation degree MR ≥ 3+);
* NYHA Classification II-IV.
* LVEF ≥ 20%
* Patients considered at high surgical risk after evaluation by two or more cardiovascular specialists (American Association for Thoracic Surgery STS score: risk of death from mitral valve repair ≥ 6% or from mitral valve replacement ≥ 8% (high risk); or the presence of 2 or more indices of frailty (moderate to severe frailty); or the presence of 2 or more major organ insufficiencies that do not improve postoperatively; or a comprehensive cardiac team assessment that the patient has other combined diseases or factors that make him or her unsuitable for surgery)
* Anatomically suitable for mitral valve repair and assessed as suitable for use of this investigational device.
* Voluntarily participate and sign an informed consent form and be willing to accept relevant examinations and clinical follow-up.

Exclusion Criteria:

* Severe mitral valve calcification
* Previous implantation of a prosthetic mitral valvuloplasty ring or prosthetic mitral valve, or previous transcatheter mitral valve surgery
* Patients with active infective endocarditis
* Patients with mitral stenosis
* Any intracardiac mass, left ventricular or atrial thrombus detected by echocardiography
* Severe coronary stenosis without surgical or interventional treatment or an acute myocardial infarction within 90 days
* Combined with tricuspid, aortic valve or severe macrovascular pathology requiring surgical or interventional treatment
* Severe pulmonary hypertension (pulmonary artery systolic pressure > 70 mmHg measured by ultrasound or right heart catheter, if measured at the same time the right heart catheter measurement shall prevail).
* Patients with severe right heart insufficiency
* Hemodynamic instability, defined as systolic blood pressure <90 mmHg in the absence of afterload-reducing drugs, cardiogenic shock, or use of intra-aortic balloon pump;
* Had a stroke/transient ischemic attack (TIA) within 30 days or severe carotid stenosis (> 70% stenosis on ultrasonography)
* Have undergone transcatheter cardiovascular intervention (PCI) within 30 days, or cardiovascular surgery within 180 days
* Have had a pacemaker or cardioverter-defibrillator (ICD) implanted, or have undergone cardiac resynchronization therapy (CRT, CRT-D) within 30 days
* Patients with clear coagulation disorders and severe coagulation disorders, or with clear contraindications to the anticoagulant drugs
* Known hypersensitivity to product composition
* Patients with severe neurological pathology affecting cognitive ability
* Patients with a life expectancy of < 12 months
* Have undergone a heart transplant or have recently been allocated a heart transplant donor
* Being enrolled in an interventional clinical study of another device or drug
* Patients diagnosed with hypertrophic cardiomyopathy, restrictive cardiomyopathy, infiltrative cardiomyopathy (e.g., amyloidosis, hemochromatosis), dilated cardiomyopathy, or constrictive pericarditis
* Patients who are pregnant or planning to become pregnant within the next 12 months. Note: Female patients of childbearing age are required to undergo a pregnancy test within 14 days prior to the operation and the result should be negative, and additionally they should use a confirmed method of contraception
* Other conditions that the investigator considers inappropriate for participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate at 12 months postoperatively | 12 months
  Clinical success is defined as no death, no mitral valve-related surgical procedures due to mitral valve incompetence, and no moderate-severe or severe mitral regurgitation (MR > 2+), with the primary evaluation indicators determined by the Core Laboratory and Clinical Event Committee (CEC).

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, Principal Investigator — FUWAI YUNAN CARDIOVASCULAR HOSPITAL

IPD SHARING:
Plan to Share IPD: No